CLINICAL TRIAL: NCT00623493
Title: Detecting Risk of Suicide in a Pediatric Emergency Department
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908070; 08-M-N070
Record Dates: First submitted 2008-02-24; First posted 2008-02-26 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05-30

CONDITIONS: Adolescents; Mental Disorder Diagnosed in Childhood; Suicide Prevention
Keywords: Screening; Suicide; Emergency Department; Children and Adolescents; Suicide Risk
MeSH Terms: conditions — Suicide Prevention; Suicide; Emergencies

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Objective:

The ultimate goal of this project is to enhance the capacity of non-mental health clinicians working in an Emergency Departments (ED) to recognize and initiate further evaluation of children and adolescents at risk for suicide.

Aim 1: To re-validate the Risk of Suicide Questionnaire (RSQ), a screening tool that assists non-psychiatric clinicians in rapidly detecting suicide risk in pediatric patients, in a pediatric ED mental health population in the Children s National Medical Center (CNMC) ED.

Aim 2: To determine the utility of a suicide screening tool, a revised version of the Risk of Suicide Questionnaire, to detect suicide risk in pediatric patients presenting to the CNMC ED for non-mental health reasons.

Study population:

The study population includes all patients admitted to the CNMC Emergency Department, ages 10 to 21, during the data collection weeks of the study period. Both patients admitted for mental health and non-mental health reasons will be included in the study.

Design:

This will be a prospective instrument development /validation study. During a designated study week, all mental health patients and a random subset of non-mental health patients admitted to the CNMC ED will be approached after their triage assessment. Following informed consent and assent, a 17-item suicide assessment tool created for this research project (RSQ-Revised), as well as a brief background questionnaire will be administered. These questions will be validated against a gold standard suicide assessment questionnaire, which will be administered to the subjects directly after the RSQ-Revised. The study aims to develop a brief suicide screening tool to be used at triage for all patients entering the ED.

Measures

Measures include the proposed 17-item screening questionnaire and a gold standard assessment of suicidal ideation in adolescents, the Suicide Ideation Questionnaire (SIQ).

DETAILED DESCRIPTION:
Objective:

The ultimate goal of this project is to enhance the capacity of non-mental health clinicians working in an Emergency Department (ED) to recognize and initiate further evaluation of children and adolescents at risk for suicide.

* Aim 1: To re-validate the Risk of Suicide Questionnaire (RSQ), a screening tool that assists non-psychiatric clinicians in rapidly detecting suicide risk in pediatric patients, in a pediatric ED mental health population.
* Aim 2: To determine the utility of a suicide screening tool, a revised version of the Risk of Suicide Questionnaire, to detect suicide risk in pediatric patients presenting to a pediatric ED for non-mental health reasons.

Study population:

This is a multi-site study and will include all patients admitted to three pediatric EDs (the Children s National Medical Center (CNMC) ED, Children s Hospital Boston (CHB) ED, and Nationwide Children s Hospital (NCH) ED), ages 10 to 21, during the data collection days of the study period. Both patients admitted for mental health and non-mental health reasons will be included in the study.

For ease of reading, from here on in, the three pediatric EDs participating in this multi-site study will be referred to as the PEDIATRIC ED.

Design:

This will be a prospective instrument development / validation study. During 5 to 10 weekdays of the month, all mental health patients and a random subset of non-mental health patients admitted to the PEDIATRIC ED will be approached after their triage assessment. Following informed consent and assent, a 17-item suicide assessment tool created for this research project (RSQ-Revised), as well as a brief background questionnaire will be administered. These questions will be validated against a gold standard suicide assessment questionnaire, which will be administered to the subjects directly after the RSQ-Revised. The study aims to develop a brief suicide screening tool to be used at triage for all patients entering the ED.

Measures

Measures include the proposed 17-item screening questionnaire and a gold standard assessment of suicidal ideation in adolescents, the Suicide Ideation Questionnaire (SIQ).

ELIGIBILITY:
* INCLUSION CRITERIA:

Patient must complete triage assessment at the PEDIATRIC ED.

For the medical patients, triage level must be 2, 3, 4 or 5, and the patient must be medically stable. For medical patients in triage level 2, in order to determine if the patient is medically stable, the interviewer will contact the ED clinician (nurse or physician) prior to approaching the patient. Any patient deemed medically unstable will not be included in the study. For the psychiatric patients, leveling is not conducted in the same way. Therefore, triage level will not be considered an exclusion factor.

Triage level in the PEDIATRIC EDs is defined by the Emergency Severity Index (ESI). ESI is a five-level ED triage algorithm that uses acuity and resource needs to stratify patients into five clinically relevant groups from 1 (most urgent) to 5 (least urgent) (Gilboy, 2005).

Age: 10-21 years.

English speaking

A legal guardian must provide informed consent and patient must sign an assent document.

EXCLUSION CRITERIA:

Developmental disability, severe cognitive impairment or communication disorder such that patient will not be able to comprehend the questions or communicate their answers

Triage level of 1 (for medical patients), indicating that the patient is not medically stable

Patient is not present with a legal guardian who can provide informed consent

Patient is non-English speaking (unfortunately, the SIQ is not available at this time in Spanish or any other languages)

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 524 (Actual)
Dates: Start 2008-02-07; Study Completion 2018-05-30

PRIMARY OUTCOMES:
Positive score on suicide assessment

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Horowitz, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (3):
- United States (3):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Childrens Hospital, Boston, Boston, Massachusetts
  - Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- [Background] Bancroft J, Hawton K, Simkin S, Kingston B, Cumming C, Whitwell D. The reasons people give for taking overdoses: a further inquiry. Br J Med Psychol. 1979 Dec;52(4):353-65. doi: 10.1111/j.2044-8341.1979.tb02536.x. PMID 508651
- [Background] Baumeister RF. Suicide as escape from self. Psychol Rev. 1990 Jan;97(1):90-113. doi: 10.1037/0033-295x.97.1.90. PMID 2408091
- [Background] Bearman PS, Moody J. Suicide and friendships among American adolescents. Am J Public Health. 2004 Jan;94(1):89-95. doi: 10.2105/ajph.94.1.89. PMID 14713704